CLINICAL TRIAL: NCT01380782
Title: Phase II Trial of Triple Receptor Tyrosine Kinase Receptor Inhibitor BIBF 1120 in Recurrent High-Grade Gliomas
Brief Title: BIBF 1120 for Recurrent High-Grade Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Y. Wen, MD (Other)
Collaborators: Boehringer Ingelheim (Industry); Wake Forest University Health Sciences (Other); University of Virginia (Other); Massachusetts General Hospital (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Patrick Y. Wen, MD, Director, Center for Neuro-Oncology, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-055; BIBF 1199.94 (Other: Boehringer-Ingleheim)
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Glioblastoma; Gliosarcoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma
Keywords: brain tumor; recurrent disease
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma; Brain Neoplasms; Recurrence | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab Naive (Experimental): Bevacizumab naive subjects
  Interventions: Drug: BIBF 1120
- Prior Bevacizumab (Experimental): Patients previously treated with bevacizumab
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120 — 200 mg BID oral for 28 day cycle

SUMMARY:
BIBF 1120 is a newly discovered compound that may stop cancer cells from growing abnormally. This drug is currently being used in treatment for other cancers in research studies and information from those other research studies suggests that this agent, BIBF 1120, may help to stop recurrent malignant glioma cells from multiplying and it may also prevent the growth of new blood vessels at the site of the tumor. In this research study, the investigators are looking to see how well BIBF 1120 works in patients with recurrent malignant gliomas.

DETAILED DESCRIPTION:
This is a two arm, multicenter, open label phase II trial in adult patients with recurrent supratentorial high-grade glioma. One arm (the "bevacizumab naïve" arm) will enroll patients who have not received prior bevacizumab therapy, and the other arm (the "post-bevacizumab" arm) will enroll patients who have experienced progression on bevacizumab.

All subjects will receive BIBF 1120 at 200mg orally, twice daily in cycles of 28 days. Subjects will come to the clinic on Day 1 of each cycle (or within 2 days prior) for blood and urine tests and a physical and neurologic exam. Bloods will also be checked within 2 days before or after Day 15 of Cycles 1 and 2. An additional blood sample will be taken on Days 1 and 8 of Cycle 1, at the start of every even-numbered cycle, and at the end of active study treatment. Subjects will have gadolinium-enhanced brain MRI scans performed with tumor measurements at screening, at the start of even-numbered cycles, and at the end of active study treatment(unless already obtained within 4 weeks of completing study treatment). 40 study subjects will have diffusion- and perfusion-weighted MRI at baseline, after 1 week on therapy (± 2 days), within 2 days prior to the start of every even-numbered cycle, and at the end of treatment (unless already obtained within 4 weeks of completing study treatment).

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically-confirmed, supratentorial, recurrent glioblastoma; subjects with an initial diagnosis of a lower grade glioma are eligible if a subsequent biopsy is determined to be glioblastoma
* Demonstration of recurrent disease on MRI following prior therapy
* Development of progressive disease after having received prior RT, and must have an interval of at least 12 weeks from the completion of any radiation therapy to study entry (unless progressive tumor growth is outside the radiation field or there is histopathological confirmation of recurrent tumor).
* Bi-dimensionally measurable disease (minimum measurement of 1 cm in one dimension) on MRI performed within 14 days prior to first treatment. (If receiving corticosteroids, participants must be on a stable or decreasing dose of corticosteroids for at least 5 days prior to baseline MRI.)
* Life expectancy of at least 12 weeks
* KPS >/= 60
* Normal organ and marrow function as defined by protocol
* Recovered from toxic effects of prior therapy
* Sufficient tumor availability (at least 15-20 unstained paraffin slides from any prior surgery)

Exclusion Criteria:

* Receiving other investigational agent
* More than 2 prior relapses
* Prior therapy with inhibitor of VEGF, VEGFR, PDGFR, or FGFR (including bevacizumab)
* Pregnant or breast-feeding
* Unwilling to agree to adequate contraception, if subject is of child-bearing potential
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BIBF 1120
* Use of EIAEDs within 14 days of registration
* Evidence of recent hemorrhage on baseline MRI of the brain
* Uncontrolled intercurrent illness
* Uncontrolled hypertension
* History of hypertensive encephalopathy
* History of any of the following within 6 months prior to enrollment: myocardial infarction or unstable angina, stroke or transient ischemic attack, significant vascular disease or peripheral arterial thrombosis, abdominal fistula, gastrointestinal perforation, or intra-abdominal abcess, intracerebral abscess
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to the first treatment day, or anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, stereotactic biopsy, fine needle aspiration, or core biopsy within 7 days prior to the first treatment day
* Serious non-healing wound, ulcer, or bone fracture
* History of a different malignancy unless disease-free for at least 5 years (unless cervical cancer in situ, or basal cell or squamous cell carcinoma of the skin)
* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wen, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Norden AD, Schiff D, Ahluwalia MS, Lesser GJ, Nayak L, Lee EQ, Rinne ML, Muzikansky A, Dietrich J, Purow B, Doherty LM, LaFrankie DC, Pulverenti JR, Rifenburg JA, Ruland SF, Smith KH, Gaffey SC, McCluskey C, Ligon KL, Reardon DA, Wen PY. Phase II trial of triple tyrosine kinase receptor inhibitor nintedanib in recurrent high-grade gliomas. J Neurooncol. 2015 Jan;121(2):297-302. doi: 10.1007/s11060-014-1631-y. Epub 2014 Oct 22. PMID 25338318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study activated at Dana-Farber Cancer Institute in May 2012 and was eventually activated at Massachusetts General Hospital, Cleveland Clinic, and University of Virginia. The bevacizumab-treated arm closed to accrual in December 2012 and the bevacizumab-naive arm closed in March 2013, both due to futility.
Groups:
- Arm A (Bevacizumab-naive) - GBM: Participants who had not been treated with bevacizumab prior to entering the study, and whose current histology was glioblastoma (GBM).
- Arm A (Bevacizumab-naive) - AG: Participants who had not been treated with bevacizumab prior to entering the study, and whose current histology was anaplastic glioma (AG).
- Arm B (Bevacizumab Treated) - GBM: Participants who had been previously treated with bevacizumab prior to entering the study, and whose currently histology was glioblastoma (GBM).
- Arm B (Bevacizumab Treated) - AG: Participants who had been previously treated with bevacizumab prior to entering the study, and whose currently histology was anaplastic glioma (AG).
Period: Overall Study
Arm/Group | Arm A (Bevacizumab-naive) - GBM | Arm A (Bevacizumab-naive) - AG | Arm B (Bevacizumab Treated) - GBM | Arm B (Bevacizumab Treated) - AG
Started | 12 | 10 | 11 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 12 | 10 | 11 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 10 | 9 | 10 | 3
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: One participant from Arm B (GBM) was removed from analysis, aside from the review of adverse events, due to later determining she did not meet eligibility requirements as a result of prior stereotatic radiosurgery received prior to starting the study.
Groups:
- Arm A Bevacizumab-naive: Bevacizumab-naive participants
- Arm B Bevacizumab-treated: Bevacizumab-treated participants
- Total: Total of all reporting groups
Arm/Group | Arm A Bevacizumab-naive | Arm B Bevacizumab-treated | Total
Number analyzed (Participants) | 22 | 14 | 36
Age, Continuous [Median (Full Range); unit: years] | 54 [28 to 75] | 52 [32 to 70] | 52 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 18
  Male | 7 | 11 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 11 | 30
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 12 | 33
  Unknown or Not Reported | 1 | 1 | 2
Karnofsky Performance Status [Median (Full Range); unit: Units on a scale] — Karnofsky Performance Status ranges from 0 (Dead) to 100 (Normal, no complaints, no evidence of disease) in increments of 10. This was measured at baseline, prior to any treatment on study.
  Units on a scale | 90 [60 to 100] | 90 [60 to 100] | 90 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: 6-Month Progression Free Survival
Description: To determine the efficacy of BIBF 1120 in bevacizumab-naive participants with recurrent glioblastoma (GBM) as measured by 6-month progression-free survival (PFS6).
Time Frame: Six months
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Bevacizumab-naive) - GBM
Number analyzed (Participants) | 12
percentage of participants | 0

2. Primary Outcome: 3-Month Progression Free Survival
Description: To determine the efficacy of BIBF 1120 in bevacizumab-treated participants with recurrent GBM as measured by 3-month progression free survival (PFS3).
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm B (Bevacizumab Treated) - GBM
Number analyzed (Participants) | 10
percentage of participants | 0

3. Secondary Outcome: Proportion of Participants Experiencing Stable Disease (SD) as Their Best Radiographic Response
Description: Best radiographic response in both populations. There were no participants with partial or complete responses, so the results are being reported in the proportion of participants who experienced stable disease (SD) as their best response (as opposed to progressive disease).
Time Frame: 2 years
Measure: Number; unit: % of patients with best response SD
Arm/Group | Arm A (Bevacizumab-naive) - GBM | Arm A (Bevacizumab-naive) - AG | Arm B (Bevacizumab Treated) - GBM | Arm B (Bevacizumab Treated) - AG
Number analyzed (Participants) | 12 | 10 | 10 | 4
% of patients with best response SD | 33 | 40 | 10 | 25

4. Secondary Outcome: Overall Survival
Description: Overall survival in both populations
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Bevacizumab-naive) - GBM | Arm A (Bevacizumab-naive) - AG | Arm B (Bevacizumab Treated) - GBM | Arm B (Bevacizumab Treated) - AG
Number analyzed (Participants) | 12 | 10 | 10 | 4
months | 6.9 [3.7 to 8.1] | 11.3 [2.7 to 14.6] | 2.6 [1.0 to 6.9] | 7.3 [1.4 to 18.1]

5. Secondary Outcome: Time-to-tumor Progression
Description: Time-to-tumor progression in both populations.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A (Bevacizumab-naive) - GBM | Arm A (Bevacizumab-naive) - AG | Arm B (Bevacizumab Treated) - GBM | Arm B (Bevacizumab Treated) - AG
Number analyzed (Participants) | 12 | 10 | 10 | 4
days | 28 [27 to 83] | 28 [27 to 138] | 28 [22 to 28] | 36 [27 to 55]

6. Secondary Outcome: Safety Profile as Summarized With Descriptive Statistics (Using Toxicity Data Gathered on Trial)
Description: Safety profile in both populations - as adverse events are posted separately in detail, these results will demonstrate serious adverse events (defined as grades 3-5) that were judged at least possibly related to Nintedanib (BIBF 1120).
Time Frame: 2 years
Measure: Number; unit: number of incidents
Arm/Group | All Participants (Arm A and B)
Number analyzed (Participants) | 37
number of incidents
  Abdominal pain | 1
  Reversible transaminase elevation | 8
  Hypertension | 1
  Hypophosphatemia | 3
  Intracranial hemorrhage | 1
  Colonic perforation | 2
  Pulmonary embolism | 1

7. Other Pre Specified Outcome: Exploratory Objective #1: Progression-free Survival at 3- and 6-months for Participants With Recurrent Anaplastic Gliomas (AG)
Description: To explore the efficacy of BIBF 1120 in bevacizumab-naïve and bevacizumab-treated participants with recurrent anaplastic gliomas (AG) survival was assessed at 6 months for Arm A and 3 months for Arm B.
Time Frame: Arm A - 6 months; Arm B - 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Bevacizumab-naive) - AG | Arm B (Bevacizumab Treated) - AG
Number analyzed (Participants) | 10 | 4
percentage of participants | 0 | 0

8. Other Pre Specified Outcome: Exploratory Objective #2: Determination if Any Correlation Exists Between Patient Outcomes (Survival, PFS3, PFS6) and Tumor Genotype and/or Expression Profile
Description: To explore the extent to which the tumor's genotype and expression profile correlate with outcome.
Time Frame: 2 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Exploratory Objective #3: Determination if Any Correlation Exists Between Patient Outcomes (Survival, PFS3, PFS6) and Serum Angiogenic Peptides, Circulating Endothelial Cells, and/or Circulating Progenitor Cells
Description: To explore the correlation between serum angiogenic peptides, circulating endothelial cells, and circulating progenitor cells with response to therapy.
Time Frame: 2 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory Objective #4: Determination if Any Correlation Exists Between Patient Outcomes (Survival, PFS3, PFS6) and Perfusion MRI, Diffusion MRI
Description: To explore the correlation between perfusion MRI, diffusion MRI and response to therapy.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected on each participant from the time the informed consent document was signed up until 30 days after the last dose of study drug.
Description: Abnormal laboratory values or diagnostic tests results constitute AEs only if they induce clinical signs or symptoms or require treatment or further diagnostic tests.
Groups:
- Arm A: Bevacizumab-naive participants
- Arm B: Bevacizumab-treated participants
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 8/22 | 5/14
Other Adverse Events (participants affected / at risk) | 22/22 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=22) | Arm B (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 3 possibly related to BIBF 1120, expected
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) — Grade 4, unrelated to BIBF 1120, unexpected
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) — Grade 3, possibly related to BIBF 1120, expected
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) — Grade 3, possibly related to BIBF 1120, expected
Colonic perforation (Gastrointestinal disorders) | 1 (2) | 0 (0) — Same participant - grade 4, possibly related to BIBF 1120 and unexpected; grade 5, possibly related to BIBF 1120 and expected.
Death NOS (General disorders) | 1 (1) | 2 (2) — Arm A - grade 5, unrelated, unexpected Arm B - both events grade 5, unrelated, unexpected
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) — Grade 3, unlikely related to BIBF 1120, unexpected
Depression (Psychiatric disorders) | 1 (1) | 0 (0) — Grade 4, unrelated to BIBF 1120, unexpected
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) — Grade 2, possibly related to BIBF 1120, unexpected
Edema cerebral (Nervous system disorders) | 1 (1) | 1 (1) — Arm A - grade 4, unlikely related to BIBF 1120, unexpected Arm B - grade <4, unrelated to BIBF 1120, unexpected
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (2) — Grade 3, unrelated to BIBF 1120, unexpected Grade 5, unrelated to BIBF 1120, unexpected
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) — Grade 3, unrelated to BIBF 1120, unexpected
Intracranial hemorrhage (Nervous system disorders) | 1 (2) | 0 (0) — Same participant - grade 2 and grade 3, possibly related to BIBF 1120, unexpected
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 2, unrelated to BIBF 1120, unexpected
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 2, possibly related to BIBF 1120, unexpected
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0) — Same participant - grade 2 twice, unrelated to BIBF 1120, and unexpected
Suicidal attempt (Psychiatric disorders) | 1 (1) | 0 (0) — Grade 3, unrelated to BIBF 1120, unexpected
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) — Arm A - grade 5, possibly related to BIBF 1120, unexpected Arm B - grade 3, unlikely related to BIBF 1120, unexpected
Vascular disorders - Other (Vascular disorders) | 0 (0) | 1 (2) — Both grade 4, one unlikely related and other unrelated to BIBF 1120, both unexpected
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=22) | Arm B (N=14)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (10) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (9) | 0 (0)
Confusion (Psychiatric disorders) | 2 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (9) | 4 (4)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Eye disorders - Other (Eye disorders) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Fatigue (General disorders) | 4 (4) | 8 (10)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 5 (6) | 6 (7)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 4 (5)
Pain (General disorders) | 1 (1) | 1 (1)
Personality change (Psychiatric disorders) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 3 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 3 (4)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3)
Weight loss (Investigations) | 2 (4) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 0 (0)
Activated partial thromboplastic time prolonged (Investigations) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 3 (3)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial intended to enroll 14 participants onto Arm A GBM, but only 10 enrolled due to futility. In addition, 10 AG participants were to be enrolled onto each Arm as exploratory cohorts, but again due to futility only 4 enrolled onto Arm B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days